CLINICAL TRIAL: NCT05605509
Title: A Phase II Study of RP-6306 in Patients With Advanced Cancer
Brief Title: RP-6306 in Patients With Advanced Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Repare Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I243
Record Dates: First submitted 2022-10-31; First posted 2022-11-04 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — Gemcitabine; IFL protocol; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- RP-6306 + Gemcitabine (Active Comparator)
  Interventions: Drug: RP-6306; Drug: Gemcitabine
- RP-6306 + FOLFIRI (Active Comparator)
  Interventions: Drug: RP-6306; Drug: FOLFIRI Protocol
- RP-6306 + Trastuzumab (Active Comparator)
  Interventions: Drug: RP-6306; Drug: Trastuzumab
- RP-6306 + RP-3500 (Active Comparator)
  Interventions: Drug: RP-6306; Drug: RP-3500

INTERVENTIONS:
Drug: RP-6306 — Dose and schedule will be assigned at enrolment
  Other Names: Lunresertib
Drug: Gemcitabine — Dose and schedule will be assigned at enrolment
  Arms: RP-6306 + Gemcitabine
Drug: FOLFIRI Protocol — Irinotecan Leucovorin FU
  Arms: RP-6306 + FOLFIRI
Drug: Trastuzumab — standard doses q3weekly
  Arms: RP-6306 + Trastuzumab
Drug: RP-3500 — Dose and schedule will be assigned at enrolment
  Other Names: Camonsertib
  Arms: RP-6306 + RP-3500

SUMMARY:
This study is being done to answer the following questions:

* Is the new drug, RP-6306, safe to use, and what effects does it have on cancer when given with standard treatment?
* If there are specific biomarkers, do patients have an improved response to treatment compared to those without the biomarker?

This study is being done to find out if this approach is better or worse than the usual approach for this type of cancer. The usual approach is defined as care most people get for this type of cancer.

DETAILED DESCRIPTION:
RP-6306 is a PKMYT1 inhibitor. PKMYT1 protein kinase negatively regulates CDK1 via phosphorylation of threonine 14 (Thr14) and sequestration in the cytoplasm. RP-6306 has shown single-agent anti-tumour efficacy in several xenograft models with amplified CCNE1 in a dose-dependent manner. RP-6306 has synergistic effects in combination with gemcitabine in CCNE1-amplified/overexpressing models in vitro and in vivo

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed cancer, that is advanced/metastatic/recurrent or unresectable, for which no curative therapy exists, and be eligible for one or more of the open cohorts
* All patients must have a formalin fixed paraffin embedded tissue block (from primary or metastatic tumour) available and must have provided informed consent for the release of the block
* Presence of clinically and/or radiologically documented disease. All radiology studies must be performed within 21 days prior to enrollment
* Patients must be ≥ 18 years of age
* Patients must have an ECOG performance status of 0 or 1
* Patients must have a life expectancy of 3 months or longer
* Hemoglobin ≥ 90 g/L (exceptions may be granted for well compensated and asymptomatic patients).
* Abs neutrophils ≥ 1.5 x 10^9/L; Platelets ≥ 100 x 10^9/L
* Bilirubin ≤ 1.5 x UNL; AST ≤2.5 x UNL; ALT ≤ 5.0 x UNL; Serum creatinine ≤ 1.5 x UNL; Creatinine clearance ≥ 50 mL/min
* Patients must be able to swallow oral medications and have no known gastrointestinal disorders that may interfere with absorption (such as malabsorption)
* Patients must have had recovered (to at least grade 0 or 1) from all reversible toxicity related to prior chemotherapy or systemic therapy and have adequate washout longest of one of the following: two weeks; 5 half-lives for investigational agents; standard cycle length of standard therapies.
* Prior external beam radiation is permitted provided a minimum of 28 days (4 weeks) have elapsed between the last dose of radiation and date of enrollment. Exceptions may be made for low-dose, non-myelosuppressive radiotherapy after consultation with CCTG. Concurrent radiotherapy is not permitted
* Previous surgery is permitted provided that a minimum of 21 days (3 weeks) have elapsed between any major surgery and date of enrollment, and that wound healing has occurred
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to screening (if applicable)/enrollment in the trial to document their willingness to participate
* Protocol treatment is to begin within 2 working days of patient enrollment
* Patients must be accessible for treatment and follow-up. Patients enrolled on this trial must be treated and followed at the participating centre
* Women/men of childbearing potential must have agreed to use a highly effective contraceptive method.

Cohort-Specific Eligibility Criteria

Cohort A: Endometrial Cancer

* Patients must have histologically confirmed diagnosis of high-grade serous endometrial cancer, that is advanced/metastatic/recurrent or unresectable, for which no curative therapy exists.
* Patients must have abnormal TP53 on IHC/genomic testing*.
* Patients must have had at least 1 prior line of platinum-based chemotherapy in any setting but may not have received prior gemcitabine therapy.

Cohort B1: HGSOC

* Patients must have a histologically confirmed diagnosis of high-grade serous ovarian cancer/fallopian tube/primary peritoneal carcinoma (HGSOC) which is platinum-refractory per standard definitions.
* Patients must have abnormal TP53 on IHC/genomic testing*.
* Platinum refractory disease refers to patients with progressive disease on first-line platinum-based chemotherapy or progressive disease within 12 weeks of the last dose of first-line platinum-based therapy [Gynecologic Cancer Intergroup Consensus Recommendations 2022].

Cohort B2: Uterine Carcinosarcoma

* Patients must have had at least 1 prior line of platinum-based chemotherapy but may not have received prior gemcitabine therapy.
* Patients must have abnormal TP53 on IHC/genomic testing*.

Cohort B3: Ovarian Carcinosarcoma

* Patients must have had at least 1 prior line of platinum-based chemotherapy but may not have received prior gemcitabine therapy.
* Patients must have abnormal TP53 on IHC/genomic testing*.

Cohort B4: TNBC

* Patients must have had at least 2 prior lines of therapy in the advanced setting.
* Patients may not have received prior gemcitabine.

Cohort B5: PDAC

* Patients must have prior FOLFIRINOX either in the palliative/advanced setting or have relapsed within 6 months of completing adjuvant or neoadjuvant FOLFIRINOX.
* Patients may not have received prior gemcitabine.
* Patients must have abnormal TP53 on IHC/genomic testing*.

Cohort B6: NSCLC

* Patients must have received standard therapies including platinum combination chemotherapy, standard salvage chemotherapy, immunotherapy, and targeted therapies as applicable.
* Patients may not have received prior gemcitabine.

Cohort C1: Colorectal Cancer

* Patients must have histologically confirmed diagnosis of colorectal cancer, that is advanced/metastatic/recurrent or unresectable, for which no curative therapy exists.
* Patients must have both a RAS mutation (KRAS) and a TP53 mutation based on local testing*.
* Patients must be eligible to receive FOLFIRI; patients homozygous for UGT1A1*28 allele are not eligible
* Patients must have had at least 1 prior line of cytotoxic chemotherapy with FOLFOX, either as:

  * 1st line therapy for metastatic disease, or
  * recurrence within 6 months of completion of adjuvant FOLFOX.

Cohort D1: HER-2+ Gastroesophageal Cancer

* Patients must have histologically confirmed diagnosis of gastroesophageal cancer, that is advanced/metastatic/recurrent or unresectable, for which no curative therapy exists.
* Tumour must be HER-2+ (IHC 3+, or FISH+) and have CCNE1 amplification

Cohort F1: Primary platinum refractory HGSOC

* Patients must have a histologically confirmed diagnosis of high grade serous ovarian cancer/fallopian tube/primary peritoneal carcinoma (HGSOC) which is platinum refractory per standard definitions.
* Patients must have one of the following for enrolment - Known CCNE1 amplification or deleterious mutations in either FBXW7 or PPP2R1A on local testing

  - Tumour designated as CCNE1 biomarker positive based on central testing (see Section 12.2)
* Platinum refractory disease refers to patients with progressive disease on first line platinum-based chemotherapy, or progressive disease within 12 weeks of the last dose of first line platinum-based therapy [Gynecologic Cancer Intergroup Consensus Recommendations 2022].

Exclusion Criteria:

* Patients with a history of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for > 2 years and which do not require ongoing treatment
* Patients with active or uncontrolled infections or with serious illnesses or medical conditions which would not permit the patient to be managed according to the protocol
* Patients are not eligible if they have a known hypersensitivity to the study drug(s) or their components
* Prior use of WEE1 inhibitor or PKMYT1 inhibitor
* Patients with significant cardiac (including uncontrolled hypertension) or pulmonary disease, or active CNS disease or infection. Patients should have a LVEF ≥ 50%.
* Patients may not receive concurrent treatment with other anti-cancer therapy (other than bone-targeted therapy, if already taking and stable) or investigational agents while on protocol therapy
* Patients who have received growth factors within 28 days prior to initiation of dosing of RP-6306 or who will require treatment with growth factors throughout the duration of the trial
* Pregnant or breastfeeding women
* Patients with history of central nervous system metastases or spinal cord compression unless they have received definitive treatment, are clinically stable and do not require corticosteroids
* Patients with any medical condition that would impair the administration of oral agents including significant bowel resection, inflammatory bowel disease or uncontrolled nausea or vomiting
* Patients who cannot discontinue the use of proton pump inhibitors, strong CYP3A inhibitors or inducers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-05-24 (Actual); Primary Completion 2025-11-14 (Actual); Study Completion 2026-02-05 (Actual)

PRIMARY OUTCOMES:
Response rate of RP-6306 in patients with selected cancers receiving standard agent | 2 years

SECONDARY OUTCOMES:
Number and severity of adverse events | 2 years
Explore the recommended dose of RP-6306 | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Lheureux, Study Chair — University Health Network, Princess Margaret Hospital, Toronto ON Canada; Yvette Drew, Study Chair — BCCA-Vancouver Cancer Centre, Vancouver BC Canada; Eric Chen, Study Chair — University Health Network, Princess Margaret Hospital, Toronto ON Canada
Locations (6):
- Canada (6):
  - BCCA - Kelowna, Kelowna, British Columbia
  - BCCA - Vancouver, Vancouver, British Columbia
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Health Sciences Centre Research Inc., London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No